CLINICAL TRIAL: NCT05425472
Title: An Open, Single-arm, Multicenter Phase II Study of HR070803 in the Treatment of Advanced Esophageal Cancer
Brief Title: A Phase II Study of HR070803 in the Treatment of Advanced Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR070803-201
Record Dates: First submitted 2022-06-01; First posted 2022-06-21 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-06

CONDITIONS: Advanced Esophageal Cancer

STUDY DESIGN:
Intervention Model Description: HR070803 for all enrolled subjects
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HR070803 (Experimental): HR070803 monotherapy will be administered by intravenous infusion
  Interventions: Drug: HR070803

INTERVENTIONS:
Drug: HR070803 — HR070803

SUMMARY:
To evaluate the efficacy, safety and pharmacokinetic characteristics of HR070803 in the treatment of advanced esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance status 0 or 1
2. Histologically confirmed advanced esophageal carcinoma
3. At least one measurable lesion is present according to the efficacy evaluation criteria for solid tumors (RECIST 1.1)
4. Able and willing to provide a written informed consent

Exclusion Criteria:

1. The tumor obviously invades adjacent organs of esophageal lesions
2. BMI≤18.5 kg/m2 or weight loss ≥10% within 2 months prior to screening
3. Subjects with unresolved adverse effects of prior therapy at the time of enrolment
4. Subjects who had received anti-tumor treatments such as surgery, chemotherapy, radiotherapy recently

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | for 4 months following the date the last patient was randomized
  The study is designed to evaluate the objective response rate of HR070803 in patients with advanced esophageal cancer. ORR is defined as percentage of patients achieving a best response of complete response (CR) or partial response (PR) as per RECIST version 1.1.

SECONDARY OUTCOMES:
Progression Free Survival | for 4 months following the date the last patient was randomized
  The study is designed to evaluate the progression free survival of HR070803 in patients with advanced esophageal cancer. PFS is defined as the time from first medication to disease progression or death, whichever is earlier
Disease Control Rate | for 4 months following the date the last patient was randomized
  The study is designed to evaluate the disease control rate of HR070803 in patients with advanced esophageal cancer. DCR is defined as the percentage of patients with a best response of CR, PR, or stable disease (SD)
Duration of Response | for 4 months following the date the last patient was randomized
  The study is designed to evaluate the duration of response of HR070803 in patients with advanced esophageal cancer. DoR is defined as the time from first documentation of response (CR or PR whichever occurred first, as per RECIST version 1.1) to disease progression or death, whichever is earlier.
Overall Survival | for 6 months following the date the last patient was randomized
  The study is designed to evaluate the overall survival of HR070803 in patients with advanced esophageal cancer. OS is defined as the time from first medication to death of any cause, censored for patients alive at data cut-off.
Number of Patients with Adverse Events as Assessed by NCI-CTCAE V5.0 | for 6 months following the date the last patient was randomized
  Safety and tolerability will consist of monitoring and recording all AEs and SAEs as characterized by type, incidence, severity, and the relationship to the study therapy. AEs will be evaluated for all treated patients using NCI-CTCAE V5.0.
ECOG Score for performance status | for 6 months following the date the last patient was randomized

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided